CLINICAL TRIAL: NCT04255966
Title: Prospective, Multi-centric, Comparative, Long-term Clinical Follow-Up Study for the Evidence of Safety and Performance Indicators of the Plasmafit® Revision Structan® Hip Endoprosthesis Cup
Brief Title: Plasmafit® Revision Structan® Hip Endoprosthesis Cup
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1821
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Osteolysis; Arthroplasty Complications; Instability of Prosthetic Joint; Degenerative Osteoarthritis; Rheumatic Arthritis; Fractures, Hip; Femoral Head Avascular Necrosis; Prosthesis Failure
Keywords: Revision of the acetabular implant; orthopaedic surgery; osteolysis; wear particles; cup loosening; malpositioned cup
MeSH Terms: conditions — Osteolysis; Joint Diseases; Rheumatic Fever; Hip Fractures; Femur Head Necrosis; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Plasmafit® Revision Structan®: Plasmafit® Revision Structan® Hip Endoprosthesis Cup
  Interventions: Device: Plasmafit® Revision Structan®

INTERVENTIONS:
Device: Plasmafit® Revision Structan® — Plasmafit® Revision Structan® Hip Endoprosthesis Cup

SUMMARY:
The aim of this observational study is to collect clinical and radiological results of the new Plasmafit® Revision Structan® Hip Endoprosthesis Cup in a standard patient population and when used in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria

* Indication for the cementless Plasmafit® Revision Structan® Hip Endoprosthesis Cup (primary and revision cases, with bone conditions typically demanding a press-fit revision cup)
* Written informed consent
* Cases where a press-fit cup fixation is possible

Exclusion Criteria

* Patients < 18 years
* Pregnant patients
* Patients not able to comply with the study demands, i.e. follow-up visits (mentally or physically)
* Patient has an infection in the hip joint region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having acute disorders of the hip, requiring primary or revision surgery, which cannot be treated by other therapies:
  * Degenerative osteoarthritis
  * Rheumatic arthritis
  * Fractures of the joint
  * Femoral head necrosis
  * Revision surgery where a sufficient intraoperative press-fit can be achieved
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (Functional results of the operated hip) over time | up to five years postoperatively
  The functional results of the operated hip will be assessed with the Harris Hip Score (HHS) and evaluated over time

SECONDARY OUTCOMES:
Survival of the implant | up to five years postoperatively
  Any removal or exchange of the acetabular cup or the polyethylene inlay is defined as revision.
  A removal of the stem is not evaluated as acetabular revision but will be documented and evaluated as part of postoperative complications.
  The revision-free survival will be assessed using the Kaplan-Meier method.
Quality of Life over time | up to five years postoperatively
  EQ-5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of three responses reflecting severity (no problems/some or moderate problems/extreme problems).
Radiological Assessment: Osseointegration of the cup over time | at 3 months, 24 months, 5 years follow-up
  The acetabular component in AP view is divided into the three regions I-III as defined by DeLee-Charnley. All three regions will be assessed for osteolysis the implant, to allow an estimation of the osseous integration and stability of the implant.
Radiological assessment: Radiographic loosening of the cup over time | at 3 months, 24 months, 5 years follow-up
  The acetabular component in AP view is divided into the three regions I-III as defined by DeLee-Charnley. All three regions will be assessed for and radiolucent lines around the implant, to allow an estimation of the osseous integration and stability of the implant.
Technical problems during surgery | Intraoperative
  Technical problems with instruments, implants or containers, instrument related issues
Impingement | Intraoperative
  The incidence of impingement during intraoperative mobilization is documented;
General handling of instruments / containers | Intraoperative
  Complaints or problems with the handling of instruments, implants or containers, instrument related issues
Complications | up to 5 years postoperatively
  All complications in the postoperative course are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Landgraeber, Prof. Dr., Principal Investigator — University Hospital, Saarland
Locations (4):
- Germany (4):
  - Orthopädische Klinik König-Ludwig-Haus, Würzburg, Bavaria
  - Herzogin Elisabeth Hospital, Braunschweig, Niedersachse
  - Gemeinschaftskrankenhaus Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland